CLINICAL TRIAL: NCT03066869
Title: Open-label, Single-center, Prospective Study on the Efficacy and Safety of Repository Corticotropin Injection (H.P. ACTHAR GEL) in the Treatment of Adults With Non-infectious Retinal Vasculitis
Brief Title: Efficacy and Safety of H.P. ACTHAR GEL in Adults With Retinal Vasculitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ocular Immunology and Uveitis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120160924
Record Dates: First submitted 2016-12-30; First posted 2017-03-01 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Uveitis, Posterior; Vasculitis Retinal
MeSH Terms: conditions — Uveitis, Posterior; Retinal Vasculitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- H.P. ACTHAR GEL (Experimental)
  Interventions: Drug: H.P. ACTHAR GEL

INTERVENTIONS:
Drug: H.P. ACTHAR GEL — H.P. Acthar Gel is an adrenocorticotropic hormone (ACTH) analogue indicated for ophthalmic diseases.

SUMMARY:
The purpose of this study is to evaluate the short- and long-term efficacy and safety of Acthar for the treatment of adults with non-infectious retinal vasculitis.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient with active retinal vasculitis (involving arteries or veins) as a manifestation of non-infectious ocular inflammatory disease; fundus must be viewable with wide-field FA in the study eye
* If both eyes are involved, both are eligible for inclusion in the study
* Patients already on non-steroidal immunosuppressive therapy may continue on this during the study, but the dose must not be increased or decreased within 6 weeks of initiating the trial
* Willing and able to sign the informed consent form

Exclusion Criteria:

* Patients under age 18
* Patients who are pregnant (must be ruled out in women of child-bearing age)
* Active infectious ocular or systemic disease
* Patients with active infectious ocular or extraocular disease
* Patients with history of malignancy, except for dermatologic entities of basal or squamous cell carcinoma which have been completely excised or removed previously
* Patients with systemic illness involving abnormalities of the hypothalamic-pituitary-adrenal axis; patients with primary adrenocortical insufficiency or adrenocortical hyperfunction
* Patients with known hypersensitivity to Acthar
* Patients on other non-steroidal systemic immunomodulatory medications with dose adjusted sooner than 6 weeks prior to study drug administration
* Patients currently on or recently treated with (within 6 weeks) systemic corticosteroid
* Patients with periocular or intraocular injections of medications administered to help control inflammation sooner than 6 weeks prior to study drug administration
* Patients with severe disease that warrants critical attention, deemed unsafe for the study by the investigator, or contraindicated, including but not limited to, patients with scleroderma, osteoporosis, systemic fungal infections, ocular herpes simplex, recent surgery, history of or the presence of a peptic ulcer, congestive heart failure, uncontrolled hypertension, or sensitivity to proteins of porcine origin. Administration of live or live attenuated vaccines is contraindicated in patients during the entire duration of the study and for one month prior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-22 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of responders to Acthar at the end of treatment. | 24 Weeks
  A responder will be defined by the binominal presence or absence of active retinal vasculitis as evaluated at Week 24. Active retinal vasculitis is defined as angiographic leakage from retinal arterioles, venules, or capillaries as determined by investigator, seen on wide-field angiography. Complete resolution or absence of active retinal vasculitis at Week 24 is considered success or "remission".

SECONDARY OUTCOMES:
Presence or absence of active retinal vasculitis at all other time points. | 1 Day to 24 Weeks
Safety assessments, including drug tolerability and adverse events; other ocular and/or systemic complications. | 1 Day to 24 Weeks
Percentage of patients requiring rescue therapy. | 1 Day to 24 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ocular Immunology & Uveitis Foundation, Waltham, Massachusetts, United States